CLINICAL TRIAL: NCT00941590
Title: Postencephalitic Symptoms After Tick Borne Encephalitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Katarina Ogrinc, University Medical Centre Ljubljana
Other Study IDs: POST-KME
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Central European Encephalitis
Keywords: tick borne encephalitis; clinical outcome; postencephalitic symptoms
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with tick borne encephalitis.

SUMMARY:
The purpose of this study is to assess clinical outcome in patients with tick borne encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* serologically proved tick borne encephalitis in patients > 15 years

Exclusion Criteria:

* pregnancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with tick borne encephalitis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Objective sequelae and subjective symptoms in patients after tick borne encephalitis. | 1 year follow-up.

SECONDARY OUTCOMES:
Comparison of subjective symptoms between patients after tick borne encephalitis and control subjects without a history of tick borne encephalitis. | 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD PhD, Study Chair — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia